CLINICAL TRIAL: NCT07275281
Title: Incidental Noncardiac Findings on Coronary Computed Tomography Angiography
Brief Title: Incidental Findings on Coronary Computed Tomography Angiography
Status: Not yet recruiting | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: JOINCIDENT.CCTA.NOV2025/3
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Computed Tomography; Coronary Angiography; Incidental Findings
Keywords: Coronary artery disease; computed tomography; indidental findings
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients who underwent CCTA: All adults (18 years of age and older0 who underwent CCTA to evaluate the coronary arteries in the past 5 years will have their CT scans reviewed for the presence of non coronary incidental findings.
  Interventions: Diagnostic Test: CCTA (Review of the scans)

INTERVENTIONS:
Diagnostic Test: CCTA (Review of the scans) — Reviewing coronary scans done in the past 5 years looking for findings other than atherosclerotic coronary artery disease.

SUMMARY:
Coronary CT angiography (CCTA) is increasingly used for ischemic heart disease diagnosis. The rising number of CCTA tests has led to a significant increase in the number of finding unexpected incidental extracardiac diseases.

DETAILED DESCRIPTION:
The increasing utilization of coronary computed tomography (CT) angiography (CCTA) to diagnose and triage patients with suspected or known ischemic heart disease has led to a parallel increase in the frequency of incidental findings in the coronaries (nonatherosclerotic), noncoronary cardiac structures and noncardiac structures.

Studies have reported a prevalence of incidental findings on CCTA up to 40%. Most of these findings have no clinical relevance, but some have significant clinical implications in the care and prognosis of the patients.

We sought to assess the frequency of incidental findings on CCTA scans in consecutive studies performed in the past 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ho underwent CCTA

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. All adult patients who underwent CCTA for chest pain diagnosis.
  2. Scans will be reviewed seeking the presence of coronary non atherosclerotic disease in the coronaries, cardiac structure and non cardiac structures.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Non atherosclerotic coronary disease | BASELINE
  Findings other than coronary atherosclerotic disease: coronary bridge, coronary dissection, coronary embolism, and coronary fistula.
Non coronary cardiac findings | BASELINE
  Findings include valve calcifications, left atrial appendage thrombus, patent foramen ovale and septal defects, pericardial effusion, LV clots, cardiac tumors.
Non cardiac findings | BASELINE
  Non cardiac findings include: a. major vascular abnormalities in the aorta and the pulmonary arteries, b. pulmonary disease: masses, lymph nodes, granulomas, and pleural effusion, and c. non pulmonary findings in the diaphragm and the hepatobiliary tree.

CONTACTS AND LOCATIONS:
Locations (1):
- Istishari Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
The excel sheet of the incidental findings in the 2000 CCTA scans in possession of the investigators will be available to any physician upon request
Supporting Information: Study Protocol, SAP